CLINICAL TRIAL: NCT04856982
Title: A Phase 3 Randomized, Placebo-Controlled Trial With a Longitudinal Natural History Run-In and Open-Label Extension to Evaluate BIIB067 Initiated in Clinically Presymptomatic Adults With a Confirmed Superoxide Dismutase 1 Mutation
Brief Title: A Study of BIIB067 (Tofersen) Initiated in Clinically Presymptomatic Adults With a Confirmed Superoxide Dismutase 1 Mutation
Acronym: ATLAS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 233AS303; 2020-004590-51 (EudraCT Number)
Expanded Access: NCT04972487 (Approved for marketing)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis Associated With a SOD1 Gene Mutation
MeSH Terms: interventions — tofersen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Natural History Run-in (No Intervention): Participants enrolled in Part A will undergo blood draws approximately once every 28 days to assess neurofilament light chain (NfL) levels.
- Part B: Randomized, Double-Blind, Placebo-Controlled (Experimental): Participants from Part A who meet the protocol-defined NfL threshold and remain presymptomatic may be eligible to participate in Part B. During Part B, participants will receive tofersen 100 milligram (mg) or placebo via intrathecal (IT) injection on Days 1, 15, 29, and every 28 days thereafter for up to approximately 5.6 years.
  Interventions: Drug: Tofersen; Drug: Placebo
- Part C: Open-Label Extension (Experimental): Participants from Part B who develop clinically manifest ALS may be eligible to participate in Part C. During Part C, participants who received placebo in Part B will receive tofersen 100 mg via IT injection on Days 1, 15, 29, and every 28 days thereafter up to the final maintenance dost visit. Participants who received tofersen during Part B will receive tofersen 100 mg on Days 1, 29, and every 28 days thereafter up to the final maintenance dost visit, with a dose of placebo on Day 15 to maintain the study blind. The combined duration of Part B and Part C is up to approximately 5.6 years.
  Interventions: Drug: Tofersen; Drug: Placebo
- Part D: Open-Label Treatment (Experimental): Participants from Part A who develop clinically manifest ALS prior to randomization in Part B may be eligible to participate in Part D. During Part D, participants will receive tofersen100 mg via IT injection on Days 1, 15, 29, and every 28 days thereafter for up to 2 years.
  Interventions: Drug: Tofersen

INTERVENTIONS:
Drug: Tofersen — Administered as specified in the treatment arm
  Other Names: BIIB067; QALSODY
  Arms: Part B: Randomized, Double-Blind, Placebo-Controlled; Part C: Open-Label Extension; Part D: Open-Label Treatment
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Part B: Randomized, Double-Blind, Placebo-Controlled; Part C: Open-Label Extension

SUMMARY:
The primary objective of this study is to evaluate the efficacy of tofersen in presymptomatic adult carriers of a superoxide dismutase 1 (SOD1) mutation with elevated neurofilament (NF). The secondary objectives of this study are to evaluate the safety and tolerability tofersen and to evaluate the effect of tofersen on pharmacodynamics (PD)/treatment response biomarkers when initiated prior to versus at the time of emergence of clinically manifest amyotrophic lateral sclerosis (ALS).

ELIGIBILITY:
Key Part A Inclusion Criteria:

* Participants should have a protocol-defined rapidly progressive SOD1 mutation, confirmed by a central reader, or a SOD1 mutation that is approved for inclusion by an external mutation adjudication committee.
* Participants with plasma NfL level less than the protocol-defined threshold.
* Participants who are clinically presymptomatic for ALS (i.e., must not have clinically manifest ALS).

Key Part A Exclusion Criteria:

* History or positive test result at screening for human immunodeficiency virus (HIV). The requirement for testing at Screening may be omitted if it is not permitted by local regulations.
* Current hepatitis C infection (defined as positive Hepatitis C Virus (HCV) antibody and detectable HCV RNA). Participants with positive HCV antibody and undetectable HCV Ribonucleic Acid (RNA) are eligible to participate in the study (United States Centers for Disease Control and Prevention).
* Current hepatitis B infection (defined as positive for hepatitis B surface antigen (HBsAg) and/or anti-Hepatitis B Core antibody (HBc)). Participants with immunity to hepatitis B from previous natural infection (defined as negative HBsAg, positive anti-HBc, and positive anti-hepatitis B surface antibody (HBs) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti- HBs) are eligible to participate in the study.
* History of systemic hypersensitivity reaction to tofersen, the excipients contained in the formulation, and if appropriate, any diagnostic agents to be administered during the study.
* History of confounding neuromuscular or neurological disorder that is expected to have a progressive (i.e., worsening) course during the study, and/or is expected to be associated with elevations in NF, in the opinion of the Investigator.
* Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that if not managed optimally could place a participant at an increased risk for intraoperative or postoperative bleeding.
* Significant cognitive impairment, clinical dementia, or unstable psychiatric illness, including psychosis, suicidal ideation, suicide attempt, or untreated major depression

  ≤ 90 days of screening, which in the opinion of the Investigator would interfere with the study procedures.
* Treatment with riluzole, edaravone, and/or sodium phenylbutyrate/taurursodiol (also known as ursodoxicoltaurine). If the participant has been on riluzole, edaravone, and/or sodium phenylbutyrate/taurursodiol, the medication(s) must be discontinued for at least 5 half-lives prior to Screening.
* Use of off-label treatments for ALS.
* Treatment with another investigational drug (including investigational drugs for ALS through compassionate use programs), biological agent, or device within 1 month or 5 half-lives of study agent, whichever is longer. Specifically, no prior treatment with small interfering RNA, stem cell therapy, or gene therapy is allowed.
* Anticipated need, in the opinion of the Investigator, for administration of any antiplatelet or anticoagulant medication (e.g., clopidogrel) that cannot be safely continued or held for an LP procedure, if necessary, according to local or institutional guidelines and/or Investigator determination.
* Current enrollment or a plan to enroll in any interventional clinical study in which an investigational treatment, biological agent, device, or approved therapy for investigational use. Participation in a noninterventional study focused on ALS natural history may be allowed at the discretion of the Investigator.

NOTE: Other protocol defined Inclusion/Exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2027-08-07 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
Parts B and C: Percentage of Participants with Emergence of Clinically Manifest ALS Within 24 Months of Part B Baseline | Up to 24 months

SECONDARY OUTCOMES:
Parts B and C: Time to Emergence of Clinically Manifest ALS | Up to 5.6 years
Parts B and C: Change in ALS Functional Rating Scale (ALSFRS-R) Total Score | Up to 5.6 years
  The ALSFRS-R measures 4 functional domains: respiratory, bulbar function, gross motor skills, and fine motor skills. There are 12 questions, each scored from 0 to 4, for a total possible score of 48, with higher scores representing better function.
Parts B and C: Change from Baseline in Percent Predicted Slow Vital Capacity (SVC) | Up to 5.6 years
Parts B and C: Percentage of Participants with Outcome as Death or Permanent Ventilation Based on Time to Death or Permanent Ventilation Analysis | Up to 5.6 years
  Permanent ventilation is defined as ≥22 hours of invasive or non-invasive mechanical ventilation per day for ≥21 consecutive days.
Parts B and C: Percentage of Participants with Outcome as Deaths Based on Time to Death Analysis | Up to 5.6 years
Parts B, C and D: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) during the Treatment Period | Parts B and C: Up to 5.6 years and Part D: Up to 2 years
Parts B, C and D: Change from Baseline in Plasma NfL Concentrations | Parts B and C: Up to 5.6 years and Part D: Up to 2 years
Parts B, C and D: Change in Total Cerebrospinal Fluid (CSF) SOD1 Concentrations | Parts B and C: Up to 5.6 years and Part D: Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (29):
- United States (12):
  - HonorHealth Neurology, Scottsdale, Arizona
  - University of California San Diego Medical Center, La Jolla, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Holy Cross Hospital Phil Smith Neuroscience Institute, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Austin Neuromuscular Center, Austin, Texas
- Macquarie University, Sydney, New South Wales, Australia
- UZ Leuven, Leuven, Flemish Brabant, Belgium
- Hospital Sao Paulo, São Paulo, São Paulo, Brazil
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Genge Partners Inc., Montreal, Quebec
- Groupe Hospitalier Pitie-Salpetriere, Paris, Paris, France
- Germany (2):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
- Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino, Italy
- Japan (2):
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - University of Tokyo Hospital, Bunkyō City, Tokyo-To
- NeuroProtect Sp. z o.o., Warsaw, Masovian Voivodeship, Poland
- Hanyang University Seoul Hospital, Seoul, South Korea
- Hospital Universitari i Politecnic La Fe, Valencia, Spain
- University Hospital of Umea, Umeå, Västerbotten County, Sweden
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Benatar M, Wuu J, Andersen PM, Bucelli RC, Andrews JA, Otto M, Farahany NA, Harrington EA, Chen W, Mitchell AA, Ferguson T, Chew S, Gedney L, Oakley S, Heo J, Chary S, Fanning L, Graham D, Sun P, Liu Y, Wong J, Fradette S. Design of a Randomized, Placebo-Controlled, Phase 3 Trial of Tofersen Initiated in Clinically Presymptomatic SOD1 Variant Carriers: the ATLAS Study. Neurotherapeutics. 2022 Jul;19(4):1248-1258. doi: 10.1007/s13311-022-01237-4. Epub 2022 May 18. PMID 35585374
- See also: Disclaimer: Residents in the United States may click here to find out more about participation in this trial. — http://www.alsATLASstudy.com